CLINICAL TRIAL: NCT01927029
Title: Prevención de Parto Prematuro en Gemelares: Ensayo Aleatorio Con Progesterona Vaginal.
Brief Title: Preterm Delivery Prevention in Twins With Progesterone
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad del Desarrollo (Other)
Collaborators: Hospital Padre Hurtado (Other); Hospital San Borja-Arriaran (Other)
Responsible Party: Principal Investigator, Masami Yamamoto, MD, Clinica Alemana de Santiago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CAS149
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Pregnancies
Keywords: twin pregnancy; progesterone; preterm delivery; >14 years; Abscense of cerclage,; TTTS, hemorrage,; history of thrombosis.; cervix >15mm
MeSH Terms: conditions — Premature Birth; Fetofetal Transfusion | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progesterone (Experimental): Daily administration of vaginal progesterone, 180mg, in gel, from 18 weeks to 34 weeks.
  Interventions: Drug: Progesterone
- Placebo (Placebo Comparator): Placebo Gel, for daily use from 18 weeks to 34 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone — Vaginal progesterone gel 180mg/daily is given from second trimester (18 to 24 weeks) until 34 weeks.
  Other Names: Progendo gel
  Arms: Progesterone
Drug: Placebo
  Arms: Placebo

SUMMARY:
Twin pregnancies have very high preterm delivery rate. Until now, no RCT has proven benefit of progesterone in this population. In contrast, singleton pregnancies are treated with this hormone. The objective is to compare 180mg/day progeterone vaginal gel with 180mg/day with placebo, from 18 weeks to 34 weeks. The sample size was calculated and 213 cases in each group are needed to demonstrate a reduction of preterm delivery <34weeks from 13% to 7%.

ELIGIBILITY:
Inclusion Criteria:

* Monochorionic or Dichorionic twin pregnancies
* 18 weeks to 24 weeks at inclusion.

Exclusion Criteria:

* Cerclage before inclusion
* Contractions, rupture of the membranes, cervix dilation,
* Short cervix (15mm or 20mm if there is history of preterm delivery
* Monoamniotic twins, Major malformation, Selective IUGR, TRAP, TTTS.
* Younger than 14 years.

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 213 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Preterm delivery <34 weeks | 14 months
  Spontaneous labor under 34 weeks.

SECONDARY OUTCOMES:
Preterm delivery <37 weeks | 14 months
  Spontaneous delivery under 37 weeks

OTHER OUTCOMES:
Neonatal mortality | 14 months
  Dead of the newborn, due to preterm delivery